CLINICAL TRIAL: NCT05951751
Title: Integrated Antenatal Screening for HIV, Syphilis, and Hepatitis B Virus (HBV) in Pregnant Women in Burkina Faso and The Gambia
Brief Title: The TRIple Elimination Model Of Mother-to-child Transmission Program (TRI-MOM)
Acronym: TRI-MOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Centre Muraz (Other); Medical Research Council (Other Government); Institut Pasteur (Industry); REVS PLUS Burkina Faso (Unknown); Young Gambian Mums Fund (Unknown); National AIDS Control Program Gambia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRD_2023_SESSTIM_TRI-MOM
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hiv; Syphilis; HBV
Keywords: maternal health; child health; HIV; Hepatitis B; Syphilis; prevention and control; pregnancy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Syphilis; Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRI-MOM (Experimental): Women attending their first postnatal visit in one of the selected maternities (no maternal age limit) will be eligible to participate in the study
  Interventions: Other: TRI-MOM intervention

INTERVENTIONS:
Other: TRI-MOM intervention — The TRI-MOM strategy includes 4 main activities:
  1. Training of healthcare professionals in charge of maternal health (nurses, midwives and doctors in charge of maternal health services)
  2. Triple screening of HIV, Syphilis and HBV by rapid diagnostic tests
  3. Assessment and treatment of women positive for any of the 3 targeted infections
  4. Raising awareness on MTCT among pregnant women visiting antenatal services and empowering women infected with at least one of the three infections

SUMMARY:
The TRI-MOM program aims to implement and evaluate a simplified (based on inexpensive rapid diagnostic tests), integrated (in governmental health facilities) and coordinated (between health care workers) strategy for the triple elimination of HIV, syphilis and HBV mother-to-child transmission (MTCT) in nine maternal and child health services, 5 in Burkina Faso and 5 in The Gambia.

The TRI-MOM program has two components:

1. an "intervention" component consisting of a pilot study to reinforce the antenatal screening and prevention of MTCT (PMTCT) capacities for the 3 targeted infections through the implementation of a simplified, integrated and coordinated strategy of triple elimination of MTCT.
2. an "evaluation" component which will assess the impact of the TRI-MOM strategy on PMTCT services, reduction of HBV MTCT and women empowerment.

DETAILED DESCRIPTION:
The TRI-MOM (TRIple elimination Model Of Mother-to-child transmission of HIV/Syphilis and HBV in Burkina Faso and The Gambia) program aims to implement and evaluate a simplified (based on inexpensive rapid diagnostic tests), integrated (in governmental health facilities) and coordinated (between health care workers) strategy for the triple elimination of HIV, syphilis and HBV MTCT in nine maternal and child health services, 5 in Burkina Faso and 5 in The Gambia. In The Gambia, the program will be conducted in collaboration with the national HIV, sexually transmitted infections (STI) and hepatitis programmes.

The TRI-MOM program has two components:

1. an "intervention" component consisting of a pilot study to reinforce the antenatal screening and PMTCT capacities for the 3 targeted infections through the implementation of a simplified, integrated and coordinated strategy of triple elimination of MTCT. This pilot study will be conducted in 9 selected maternities.
2. an "evaluation" component which will assess the impact of the TRI-MOM strategy on PMTCT services, reduction of HBV MTCT and women empowerment.

Intervention component :

The TRI-MOM strategy includes 4 main activities:

1. Training of healthcare professionals in charge of maternal health (nurses, midwives and doctors in charge of maternal health services)
2. Triple screening of HIV, Syphilis and HBV by rapid diagnostic tests
3. Assessment and treatment of women positive for any of the 3 targeted infections
4. Raising awareness on MTCT among pregnant women visiting antenatal services and empowering women infected with at least one of the three infections

Evaluation component :

The TRI-MOM program will include three studies :

1. A quantitative and qualitative cross-sectional study before and after the implementation of the strategy.
2. A cohort study of pregnant women positive for any of the three infections.
3. Cost and cost-effectiveness analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women attending a postnatal visit in one of the selected maternities (no maternal age limit)

Exclusion Criteria:

* Refusal to participate in the study
* Unable to provide consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Coverage of the strategy in the study maternities before its implementation | Assessed cross-sectionally using a questionnaire administered to women at baseline (before the implementation of the TRI-MOM strategy)
  Proportion of women screened for HIV, Syphilis and HBV during pregnancy
Coverage of the strategy in the study maternities after its implementation | Assessed cross-sectionally using a questionnaire administered to women at 12 months (after the implementation of the TRI-MOM strategy)
  Proportion of women screened for HIV, Syphilis and HBV during pregnancy

SECONDARY OUTCOMES:
Knowledge of the targeted infections before the strategy implementation | Assessed cross-sectionally using a questionnaire administered to women at baseline (before the implementation of the TRI-MOM strategy)
  Proportion of women with a good level of knowledge (defined by a score) of the targeted infections (HIV, syphilis, and HBV) and of PMTCT
Knowledge of the targeted infections after the strategy implementation | Assessed cross-sectionally using a questionnaire administered to women at 12 months (after the implementation of the TRI-MOM strategy)
  Proportion of women with a good level of knowledge (defined by a score) of the targeted infections (HIV, syphilis, and HBV) and of PMTCT
Acceptability of the implemented strategy and PMTCT and preferences : screening refusal before the strategy implementation | Assessed cross-sectionally using a questionnaire administered to women at baseline (before the implementation of the TRI-MOM strategy)
  Proportion of pregnant women who refuse the screening for any of the 3 targeted infections
Acceptability of the implemented strategy and PMTCT and preferences : screening refusal after the strategy implementation | Assessed cross-sectionally using a questionnaire administered to women at 12 months (after the implementation of the TRI-MOM strategy)
  Proportion of pregnant women who refuse the screening for any of the 3 targeted infections
Acceptability of the implemented strategy and PMTCT and preferences : treatment refusal before the strategy implementation | Assessed cross-sectionally using a questionnaire administered to women at baseline (before the implementation of the TRI-MOM strategy)
  Proportion of positive pregnant women refusing treatment
Acceptability of the implemented strategy and PMTCT and preferences : treatment refusal after the strategy implementation | Assessed cross-sectionally using a questionnaire administered to women at 12 months (after the implementation of the TRI-MOM strategy)
  Proportion of positive pregnant women refusing treatment
Sensitivity of the hepatitis B core-related antigen rapid diagnostic test (HBcrAg-RDT) (PROTECT-B ancillary study) | Data collected at cohort inclusion
  Percentage of HBsAg-positive women with a high viral load (≥200,000 IU/mL) who are positive for HBcrAg-RDT
Specificity of the HBcrAg-RDT (PROTECT-B ancillary study) | Data collected at cohort inclusion
  Percentage of HBsAg-positive women with a low viral load <200,000 IU/mL who are negative for HBcrAg-RDT
Positive predictive value of the HBcrAg-RDT (PROTECT-B ancillary study) | Data collected at cohort inclusion
  Proportion of subjects with a positive HBcrAg test result who truly have a high viral load (≥200,000 IU/mL)
Negative predictive value of the HBcrAg-RDT (PROTECT-B ancillary study) | Data collected at cohort inclusion
  Proportion of subjects with a negative HBcrAg test result who truly do not have a high viral load (≥200,000 IU/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Boyer, PhD, Principal Investigator — UMR 1252 SESSTIM
Locations (2):
- Centre Muraz/INSP, Bobo-Dioulasso, Burkina Faso
- MRC The Gambia at LSHTM, Fajara, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
To be completed

REFERENCES:
- [Derived] Vo-Quang E, Guingane AN, Perieres L, Ndow G, Some V, Badjie S, Jobe A, Gouem C, Shimakawa Y, Kania D, Lemoine M, Boyer S; TRI-MOM study group. Towards triple elimination of HIV, syphilis and HBV mother-to-child transmission: Protocol of a simplified and integrated strategy in Burkina Faso and The Gambia: Protocol for the phase 1 of the TRI-MOM project. PLoS One. 2026 Feb 6;21(2):e0322670. doi: 10.1371/journal.pone.0322670. eCollection 2026. PMID 41649980